CLINICAL TRIAL: NCT04002063
Title: Does Adding a Tailored Cognitive Behavioral Therapy (CBT) Mobile Skills App Mediate Higher Rates of Depression Recovery, Adjustment, and Quality of Life in OEF/OIF Veterans Compared to Standard CBT?
Brief Title: Does Adding a Tailored Cognitive Behavioral Therapy (CBT) Mobile Skills App Mediate Rates of Depression
Acronym: CBTMobileV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2908-R
Record Dates: First submitted 2019-06-20; First posted 2019-06-28 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Depression
Keywords: Depression; OEF/OIF; Mobile Apps; Cognitive Behavioral Therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: a full-scale multi-site randomized clinical trial (RCT) to measure the efficacy of CBT-D enhanced with CBT MobileWork-V, a comprehensive CBT skill training smartphone app (the experimental arm) for improving CBT understanding and skill acquisition and depressive symptoms, in OEF/OIF Veterans with depression compared to standard CBT-D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT-D augmented with CBT MobileWork-V (Experimental): Patients randomized to this condition will receive CBT-D as usual plus access to CBT MobileWork-V, a comprehensive tailored smartphone app for CBT skills practice for OEF/OIF Veterans.
  Interventions: Behavioral: CBT MobileWork-V plus CBT
- CBT-D (Active Comparator): Patients randomized to CBT-D will receive CBT-D as usual only.
  Interventions: Behavioral: CBT MobileWork-V plus CBT; Behavioral: CBT alone

INTERVENTIONS:
Behavioral: CBT MobileWork-V plus CBT — a smartphone app to assist with CBT homework skills practice plus CBT
Behavioral: CBT alone — CBT therapy individual
  Other Names: CBT-D
  Arms: CBT-D

SUMMARY:
Depression is a common psychological disorder seen in 18.5% of Operation Enduring Freedom (OEF), Operation Iraqi Freedom (OIF), and Operation New Dawn (OND) Veterans. Improving the rate of depression recovery and remission is vital to enhance OEF/OIF/OND Veteran's ability to improve work and home adjustment and overall quality of life. OEF/OIF/OND Veterans have reported many barriers to following through with Cognitive therapy skills practice assignments, a key component of CBT therapy, the leading therapy for depression in the VA. Smartphone apps have been identified as a useful widely-used tool to improve the effectiveness of psychological treatments. The investigators propose a full-scale multi-site randomized clinical trial (RCT) to measure the efficacy of CBT-D enhanced with CBT MobileWork-V, a comprehensive CBT skill training smartphone app (the experimental arm) for improving CBT understanding and skill acquisition and depressive symptoms, in OEF/OIF Veterans with depression compared to standard CBT-D.

DETAILED DESCRIPTION:
Cognitive Behavioral Therapy (CBT) is the leading evidence-based psychotherapy for depression, which affects 18.5% of Operation Enduring Freedom (OEF), Operation Iraqi Freedom (OIF), and Operation New Dawn (OND) Veterans (hereafter referred to as OEF/OIF). Yet, OEF/OIF Veterans had only a 30% average reduction in mean depression scores from the initial to later phase of treatment. This was true despite the rigorous training and certification procedures for VA CBT-D. Improving the rate of depression recovery and remission is vital to enhance OEF/OIF Veteran's ability to improve work and home adjustment and overall quality of life.

Broad access to all key ingredients of CBT, including skills practice (homework), is associated with improved and faster recovery from depression. OEF/OIF Veterans and patients with depression have reported many barriers (i.e., time, chaotic lifestyles, and low energy) to following through with their skills practice assignments. In the absence of targeted strategies/interventions to address the barriers that prevent CBT skills practice, OEF/OIF Veterans will remain unable to reap the full benefits/effects of CBT. With specific tailored interventions to address this gap in treatment, OEF/OIF Veterans will improve rates of recovery from depression, diminished home and work adjustment, and poor quality of life.

Leveraging the technological savvy of this generation of Veterans to improve access to CBT skills practice is a logical tactic to address this gap in treatment. Smartphone apps have been identified as a useful widely-used tool to improve the effectiveness of psychological treatments. There is, however, a paucity of empirical studies on the use of mobile apps in the treatment of depressed OEF/OIF Veterans and in psychological treatment overall. The promising pilot results of a comprehensive tailored smartphone app for CBT skills practice for OEF/OIF Veterans ("CBT MobileWork-V"), provides initial evidence for a larger-scale randomized clinical trial (RCT) to measure the efficacy of CBT enhanced with CBTMobileWork-V (the experimental arm) for improving CBT understanding and skill acquisition and depressive symptoms, in OEF/OIF Veterans with depression compared to standard CBT-D. Specifically, over a 27-month period the study will randomize 268 eligible OEF/OIF Veterans with depressive symptoms, to either CBT augmented with the comprehensive CBT skill training smartphone app CBT MobileWork-V or standard CBT-D with traditional skills practice methods (i.e., paper and pencil). The Specific Aims of this study are:

Primary Aim 1) To assess whether CBT-D augmented with CBT MobileWork-V (hereafter referred to as CBT-D+) promotes greater CBT understanding and skill acquisition compared to traditional CBT-D.

Primary Aim 2a) To examine the short-term effect in depressive symptoms after 12 weeks of CBT-D+ versus standard CBT-D.

Primary Aim 2b) To examine the long-term effect in depressive symptoms at 6 months post treatment of the CBT-D+ intervention versus traditional CBT-D.

ELIGIBILITY:
Inclusion Criteria:

* Veteran of OEF/OIF/OND deployments
* Depressive severity of at least 10 on the PHQ-9 at screening (Patient may also have a DSM-5 56 diagnosis of unipolar Major Depression; PTSD; any anxiety disorder; substance/alcohol abuse; or adjustment disorder)
* Ability to read at the eighth grade level and to provide informed consent
* Patients may be taking antidepressants or antianxiety medications where dose has been stable for at least 4 weeks prior to screening evaluation
* Must have an Android smartphone
* Must be willing to be audio-taped for fidelity ratings

Exclusion Criteria:

* Diagnoses of schizophrenia, schizo-affective, bipolar, or other psychotic disorder
* Serious suicidal risk (Patient responds positively to PHQ-9 question #9) See B.3.4.1.
* Severe PTSD (Score greater than 51 on PTSD Checklist for DSM-5)
* Severe substance or alcohol dependence (meets DSM-5 criteria of severe)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Ann Callan, PhD RN, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (9):
- United States (9):
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Rehabilitation R&D Service, Baltimore, MD, Baltimore, Maryland
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Coatesville VA Medical Center, Coatesville, PA, Coatesville, Pennsylvania
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CBT-D Augmented With CBT MobileWork-V | CBT-D
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT-D Augmented With CBT MobileWork-V | CBT-D | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
PHQ-9 [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire-9 (PHQ-9) is a screening tool for assessing depression.It is a self-reported questionnaire that helps gauge the severity of depressive symptoms.
  Components of PHQ-9
  . Each question asks the patient to rate how often they have been bothered by specific problems over the past two weeks.
  Interpreting PHQ-9 Scores The total score on the PHQ-9 ranges from 0 to 27.
  * 0-4: Minimal or no depression
  * 5-9: Mild depression
  * 10-14: Moderate depression
  * 15-19: Moderately severe depression
  * 20-27: Severe depression
  units on a scale | 15.629 (2.004) | 20.915 (1.814) | 17.352 (1.603)
Dimensions of Anger Reactions [Mean (Standard Deviation); unit: units on a scale] — The Dimensions of Anger Reactions Scale (DAR-5) looks at anger over the previous 4 weeks including the frequency, intensity, duration, level of aggression and impact on functioning. It has been validated in Australian populations and is a useful and quick way to assess problematic anger. You will get a total severity score (range 5-25). Higher scores indicate more symptoms and a score above 12 indicates that you are experiencing psychological distress and functional impairment as a result of anger.
  units on a scale | 11.595 (.843) | 12.298 (.970) | 11.946 (.643)
GAD [Mean (Standard Deviation); unit: units on a scale] — The Generlized Anxiety Scale (GAD-7) is a widely used self-administered screening tool for Generalized Anxiety Disorder (GAD), designed to assess the severity of anxiety symptoms over the past two weeks.
  days The total score can range from 0 to 21. Higher scores indicate greater severity of anxiety symptoms.
  Interpretation of Scores 0-4: Minimal anxiety 5-9: Mild anxiety 10-14: Moderate anxiety 15-21: Severe anxiety A score of 10 or greater is often used as a threshold for further evaluation, indicating a higher likelihood of GAD.
  units on a scale | 21.064 (1.415) | 17.913 (1.671) | 19.489 (1.095)
PTSD Checklist [Mean (Standard Deviation); unit: units on a scale] — The Posttraumatic Stress Disorder (PTSD) Checklist is known as the PCL, it is a self-screening tool to help in the diagnosis of PTSD. The score is worked out by adding up the number of points for each answer. The minimum score is 0, the maximum is 80. In addition, a score of 38 or higher indicates probable PTSD in veterans; the score may be set higher or lower for civilians; no agreement has been reached yet since it was only developed after the DSM-5 was published in 2013.
  units on a scale | 55.488 (4.282) | 48.022 (5.203) | 51.755 (3.369)
Military to Civilian Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Military to Civilian Questionnaire (M2C-Q) is a brief 16-item self-report measure of postemployment reintegration difficulty among veterans. Items are rated on a 5-point likert scale ranging from 0 = no difficulty to 4 = extreme difficulty. Higher scores indicate greater postemployment difficulty. Scores range from 0 to 64, with higher scores indicating greater difficulty with post deployment integration.
  units on a scale | 55.230 (3.093) | 52.608 (1.830) | 53.919 (1.797)
Quality of Life Questionnaire [Mean (Standard Deviation); unit: units on a scale] — WHOQOL stands for the World Health Organization Quality of Life assessment which measures quality of life across different cultures. It assesses individuals' perceptions of their health and well-being, taking into account various domains of life: physical health, psychological state, social relationships, and environment. WHOQOL (total score 0-100) uses a 5-point Likert scale, where participants rate their responses from 1 to 5, with higher scores indicating better quality of life. The data are scored to yield an overall quality of life score, as well as sub-scores for each of the six domains.
  units on a scale | 77.205 (4.016) | 79.182 (2.875) | 78.194 (2.470)

OUTCOME MEASURES:

1. Primary Outcome: Skills of Cognitive Therapy (Patient Version)
Description: The Skills of Cognitive Therapy Scale (SoCT) is 8-item self-report (patient version) of a 5-point Likert-type scale ranging from 1 (never) to 5 (always or when needed) assesses patients understanding and use of basic CBT skills in depressed adults. The eight-item SoCT assesses patients' understanding and use of basic cognitive therapy (CT) skills rated from the perspectives of patients (SoCT-P). Ratings of patients' skill usage are made on 5-point Likert-type scales ranging from 1 ("never") to 5 ("always or when needed"). Total scores range 8 - 40. Higher scores reflect greater patient skill in applying cognitive therapy principles and coping strategies.
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT-D Augmented With CBT MobileWork-V | CBT-D
Number analyzed (Participants) | 8 | 7
units on a scale | 24.231 (1.495) | 24.231 (1.495)

2. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire-9 (PHQ-9) is a screening tool for assessing depression. It is a self-reported questionnaire that helps gauge the severity of depressive symptoms. Components of PHQ-9. Each question asks the patient to rate how often they have been bothered by specific problems over the past two weeks. The total score on the PHQ-9 ranges from 0 to 27.
  Interpreting PHQ-9 Scores:
  0-4: Minimal or no depression 5-9: Mild depression 10-14: Moderate depression 15-19: Moderately severe depression 20-27: Severe depression
Time Frame: week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CBT-D Augmented With CBT MobileWork-V | CBT-D
Number analyzed (Participants) | 8 | 7
units on a scale | 23.798 [19.680 to 27.916] | 18.004 [13.082 to 22.926]

ADVERSE EVENTS:
Time Frame: up to 24 weeks
Description: No adverse events
Arm/Group | CBT-D Augmented With CBT MobileWork-V | CBT-D
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

LIMITATIONS AND CAVEATS:
* COVID 19 pandemic & Contracts for s/w programmers delayed, Programming & bug fixes from prototype, enhanced features, & Veteran specific materials
* Contract for data server & website at the U Pittsburgh delayed, VA cyber security approval (2.5 years), Admin delays, especially during COVID)- CIRB, staff onboarding, site onboarding, local sites IRB, Therapist onboarding delays: VAMC clinician shortages, Trends in CBT treatment (less visits, group therapy, etc.) changed since study inception

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT04002063/Prot_SAP_001.pdf